CLINICAL TRIAL: NCT01477476
Title: Anti-IL-1 Treatment in Children Diabetic Keto-Acidosis (DKA) at Diagnosis of Type 1 Diabetes.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: funding loss, no data was ever collected
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-0814; P30DK057516 (NIH)
Record Dates: First submitted 2011-11-18; First posted 2011-11-22 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Type I Diabetes
Keywords: DKA; Diabetes; Type I Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Treatment (Active Comparator): 14 subjects with receive active treatment with Anakinra.
  Interventions: Drug: Anakinra
- Placebo (Placebo Comparator): 7 subjects will receive the placebo comparator.
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Drug: Anakinra — Anakinra treatment will be given I.V. as a bolus of 2 mg/kg infused intravenously over 30 minutes followed by infusion of 2 mg/kg/hour for 4 hours.
  Other Names: anti Interleukin 1 receptor antibodies
  Arms: Active Treatment
Other: Placebo Comparator — A placebo will be given to 7 subjects.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled phase 2 study. Specific aim is to evaluate feasibility and safety of anti-IL-1 (interleukin 1) treatment in the course of standard therapy for diabetic ketoacidosis in children and its effect on intracranial pressure.

DETAILED DESCRIPTION:
Anakinra is a fully human IL-1ra (interleukin 1 receptor agonist) licensed in 2001 by FDA for the treatment of rheumatoid arthritis. It competitively binds to the IL-1 receptor, thus blocking IL-1 signaling. It is a short-acting agent that requires daily subcutaneous administration at 1-2 mg/kg, maximum 100 mg/dose. It has been effective in lowering HbA1c (glycated haemoglobin) in T2D (type 2 diabetes) and a randomized trial of anakinra in recent onset T1D (type 1 diabetes) is underway in Europe. Overall, anakinra has been used in adults and children with a good safety record, for more than 10 years. Infrequent side effects include infections, neutropenia, nausea, diarrhea, cardiopulmonary arrest, influenza-like symptoms, and production of anti-anakinra antibodies.

Study Design: A double-blinded placebo-controlled RCT (randomized controlled trial) with 2:1 allocation (14 active treatment vs. 7 placebo). Anakinra treatment will be given as a bolus of 2 mg/kg infused intravenously over 30 minutes followed by infusion of 2 mg/kg/hour for 4 hours immediately after confirmation of the diagnosis of DKA (diabetic keto-acidosis) and when laboratory safety parameters are available (CBC (complete blood count) and pregnancy test) and after a consent is obtained. Primary outcomes: Safety and tolerability of anti-IL-1 treatment (anakinra) during the initial 24 hr period of DKA treatment. Secondary outcomes: Optic nerve sheath diameter (cut-off to define cerebral edema: 4.5 mm); Changes in cytokines levels during the treatment with anakinra.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-18 years at diagnosis of type 1 diabetes
* Diabetic ketoacidosis with:

  * plasma glucose concentration >300 mg/dl,
  * venous pH <7.30 or
  * serum bicarbonate concentration <15 mmol/L, and
  * ketones in urine or serum
* Hematology:

  * WBC >3000 x 109/L;
  * platelets >100,000 x 109/L;
  * hemoglobin >10.0 g/dL
* Negative blood pregnancy test in females.

Exclusion Criteria:

* Children with underlying disorders, including:

  * active autoimmune or immune deficiency disorder other than type 1 diabetes,
  * malignancy,
  * organ transplant,
  * any condition requiring chronic corticosteroid use
* Previous immunotherapy to prevent type 1 diabetes
* Current or prior infection with HIV, hepatitis B or hepatitis C assessed by history
* Patients who present with DKA concomitant with alcohol or drug use,
* Head trauma,
* Meningitis or other conditions which might affect neurological function
* Renal failure
* Any condition, medical or otherwise that would, in the opinion of the investigator, prevent complete participation in the study, or that would pose a significant hazard to the subject's participation
* Patients with a history of known hypersensitivity to:

  * E coli-derived proteins,
  * anakinra, or
  * any components of the investigational drug product

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-04-22 (Actual)

PRIMARY OUTCOMES:
Frequency of Adverse Events | 24 hours
  Type and number of Adverse Events related to anti-IL-1 treatment (anakinra) during the initial 24 hour period of DKA treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Arleta Rewers, MD, Phd, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - Childrens Hospital Colorado, Aurora, Colorado
  - University of Colorado, Anschutz Medical Campus, Aurora, Colorado

REFERENCES:
- [Background] Rewers A, Chase HP, Mackenzie T, Walravens P, Roback M, Rewers M, Hamman RF, Klingensmith G. Predictors of acute complications in children with type 1 diabetes. JAMA. 2002 May 15;287(19):2511-8. doi: 10.1001/jama.287.19.2511. PMID 12020331
- [Background] Rewers A, Klingensmith G, Davis C, Petitti DB, Pihoker C, Rodriguez B, Schwartz ID, Imperatore G, Williams D, Dolan LM, Dabelea D. Presence of diabetic ketoacidosis at diagnosis of diabetes mellitus in youth: the Search for Diabetes in Youth Study. Pediatrics. 2008 May;121(5):e1258-66. doi: 10.1542/peds.2007-1105. PMID 18450868
- [Background] Maniatis AK, Goehrig SH, Gao D, Rewers A, Walravens P, Klingensmith GJ. Increased incidence and severity of diabetic ketoacidosis among uninsured children with newly diagnosed type 1 diabetes mellitus. Pediatr Diabetes. 2005 Jun;6(2):79-83. doi: 10.1111/j.1399-543X.2005.00096.x. PMID 15963034
- [Background] Muir AB, Quisling RG, Yang MC, Rosenbloom AL. Cerebral edema in childhood diabetic ketoacidosis: natural history, radiographic findings, and early identification. Diabetes Care. 2004 Jul;27(7):1541-6. doi: 10.2337/diacare.27.7.1541. PMID 15220225
- [Background] Glaser NS, Wootton-Gorges SL, Buonocore MH, Marcin JP, Rewers A, Strain J, DiCarlo J, Neely EK, Barnes P, Kuppermann N. Frequency of sub-clinical cerebral edema in children with diabetic ketoacidosis. Pediatr Diabetes. 2006 Apr;7(2):75-80. doi: 10.1111/j.1399-543X.2006.00156.x. PMID 16629712
- [Background] Edge JA, Hawkins MM, Winter DL, Dunger DB. The risk and outcome of cerebral oedema developing during diabetic ketoacidosis. Arch Dis Child. 2001 Jul;85(1):16-22. doi: 10.1136/adc.85.1.16. PMID 11420189
- [Background] Edge JA. Cerebral oedema during treatment of diabetic ketoacidosis: are we any nearer finding a cause? Diabetes Metab Res Rev. 2000 Sep-Oct;16(5):316-24. doi: 10.1002/1520-7560(2000)9999:99993.0.co;2-r. PMID 11025556
- [Background] Glaser N, Barnett P, McCaslin I, Nelson D, Trainor J, Louie J, Kaufman F, Quayle K, Roback M, Malley R, Kuppermann N; Pediatric Emergency Medicine Collaborative Research Committee of the American Academy of Pediatrics. Risk factors for cerebral edema in children with diabetic ketoacidosis. The Pediatric Emergency Medicine Collaborative Research Committee of the American Academy of Pediatrics. N Engl J Med. 2001 Jan 25;344(4):264-9. doi: 10.1056/NEJM200101253440404. PMID 11172153
- [Background] Wolfsdorf J, Glaser N, Sperling MA; American Diabetes Association. Diabetic ketoacidosis in infants, children, and adolescents: A consensus statement from the American Diabetes Association. Diabetes Care. 2006 May;29(5):1150-9. doi: 10.2337/diacare.2951150. No abstract available. PMID 16644656
- [Background] Blamire AM, Anthony DC, Rajagopalan B, Sibson NR, Perry VH, Styles P. Interleukin-1beta -induced changes in blood-brain barrier permeability, apparent diffusion coefficient, and cerebral blood volume in the rat brain: a magnetic resonance study. J Neurosci. 2000 Nov 1;20(21):8153-9. doi: 10.1523/JNEUROSCI.20-21-08153.2000. PMID 11050138
- [Background] Hoffman WH, Burek CL, Waller JL, Fisher LE, Khichi M, Mellick LB. Cytokine response to diabetic ketoacidosis and its treatment. Clin Immunol. 2003 Sep;108(3):175-81. doi: 10.1016/s1521-6616(03)00144-x. PMID 14499240
- [Background] Glaser N. Cerebral injury and cerebral edema in children with diabetic ketoacidosis: could cerebral ischemia and reperfusion injury be involved? Pediatr Diabetes. 2009 Dec;10(8):534-41. doi: 10.1111/j.1399-5448.2009.00511.x. Epub 2009 Oct 10. No abstract available. PMID 19821944
- [Background] Mulcahy NJ, Ross J, Rothwell NJ, Loddick SA. Delayed administration of interleukin-1 receptor antagonist protects against transient cerebral ischaemia in the rat. Br J Pharmacol. 2003 Oct;140(3):471-6. doi: 10.1038/sj.bjp.0705462. Epub 2003 Aug 26. PMID 12970087
- [Background] Banwell V, Sena ES, Macleod MR. Systematic review and stratified meta-analysis of the efficacy of interleukin-1 receptor antagonist in animal models of stroke. J Stroke Cerebrovasc Dis. 2009 Jul-Aug;18(4):269-76. doi: 10.1016/j.jstrokecerebrovasdis.2008.11.009. PMID 19560680
- [Background] Clark SR, McMahon CJ, Gueorguieva I, Rowland M, Scarth S, Georgiou R, Tyrrell PJ, Hopkins SJ, Rothwell NJ. Interleukin-1 receptor antagonist penetrates human brain at experimentally therapeutic concentrations. J Cereb Blood Flow Metab. 2008 Feb;28(2):387-94. doi: 10.1038/sj.jcbfm.9600537. Epub 2007 Aug 8. PMID 17684519
- [Background] Emsley HC, Smith CJ, Georgiou RF, Vail A, Hopkins SJ, Rothwell NJ, Tyrrell PJ; Acute Stroke Investigators. A randomised phase II study of interleukin-1 receptor antagonist in acute stroke patients. J Neurol Neurosurg Psychiatry. 2005 Oct;76(10):1366-72. doi: 10.1136/jnnp.2004.054882. PMID 16170078
- [Background] Leslie KS, Lachmann HJ, Bruning E, McGrath JA, Bybee A, Gallimore JR, Roberts PF, Woo P, Grattan CE, Hawkins PN. Phenotype, genotype, and sustained response to anakinra in 22 patients with autoinflammatory disease associated with CIAS-1/NALP3 mutations. Arch Dermatol. 2006 Dec;142(12):1591-7. doi: 10.1001/archderm.142.12.1591. PMID 17178985
- [Background] Lachmann HJ, Kone-Paut I, Kuemmerle-Deschner JB, Leslie KS, Hachulla E, Quartier P, Gitton X, Widmer A, Patel N, Hawkins PN; Canakinumab in CAPS Study Group. Use of canakinumab in the cryopyrin-associated periodic syndrome. N Engl J Med. 2009 Jun 4;360(23):2416-25. doi: 10.1056/NEJMoa0810787. PMID 19494217
- [Background] Kitley JL, Lachmann HJ, Pinto A, Ginsberg L. Neurologic manifestations of the cryopyrin-associated periodic syndrome. Neurology. 2010 Apr 20;74(16):1267-70. doi: 10.1212/WNL.0b013e3181d9ed69. PMID 20404307
- [Background] Mandrup-Poulsen T, Bendtzen K, Nerup J, Dinarello CA, Svenson M, Nielsen JH. Affinity-purified human interleukin I is cytotoxic to isolated islets of Langerhans. Diabetologia. 1986 Jan;29(1):63-7. doi: 10.1007/BF02427283. PMID 3514344
- [Background] Atkinson MA, Wilson SB. Fatal attraction: chemokines and type 1 diabetes. J Clin Invest. 2002 Dec;110(11):1611-3. doi: 10.1172/JCI17311. No abstract available. PMID 12464665
- [Background] Mandrup-Poulsen T, Pickersgill L, Donath MY. Blockade of interleukin 1 in type 1 diabetes mellitus. Nat Rev Endocrinol. 2010 Mar;6(3):158-66. doi: 10.1038/nrendo.2009.271. PMID 20173777
- [Background] Kaas A, Pfleger C, Hansen L, Buschard K, Schloot NC, Roep BO, Mortensen HB; Hvidore Study Group on Childhood Diabetes. Association of adiponectin, interleukin (IL)-1ra, inducible protein 10, IL-6 and number of islet autoantibodies with progression patterns of type 1 diabetes the first year after diagnosis. Clin Exp Immunol. 2010 Sep;161(3):444-52. doi: 10.1111/j.1365-2249.2010.04193.x. PMID 20529086
- [Background] Pickersgill LM, Mandrup-Poulsen TR. The anti-interleukin-1 in type 1 diabetes action trial--background and rationale. Diabetes Metab Res Rev. 2009 May;25(4):321-4. doi: 10.1002/dmrr.960. PMID 19405081
- [Background] Kindt S, Vanden Berghe P, Boesmans W, Roosen L, Tack J. Prolonged IL-1beta exposure alters neurotransmitter and electrically induced Ca(2+) responses in the myenteric plexus. Neurogastroenterol Motil. 2010 Mar;22(3):321-e85. doi: 10.1111/j.1365-2982.2009.01414.x. Epub 2009 Oct 1. PMID 19796332
- [Background] Schroder K, Zhou R, Tschopp J. The NLRP3 inflammasome: a sensor for metabolic danger? Science. 2010 Jan 15;327(5963):296-300. doi: 10.1126/science.1184003. PMID 20075245
- [Background] Larsen CM, Faulenbach M, Vaag A, Volund A, Ehses JA, Seifert B, Mandrup-Poulsen T, Donath MY. Interleukin-1-receptor antagonist in type 2 diabetes mellitus. N Engl J Med. 2007 Apr 12;356(15):1517-26. doi: 10.1056/NEJMoa065213. PMID 17429083
- [Background] Larsen CM, Faulenbach M, Vaag A, Ehses JA, Donath MY, Mandrup-Poulsen T. Sustained effects of interleukin-1 receptor antagonist treatment in type 2 diabetes. Diabetes Care. 2009 Sep;32(9):1663-8. doi: 10.2337/dc09-0533. Epub 2009 Jun 19. PMID 19542207
- [Background] Donath, M. Y., Weder, C., and Brunner, A. XOMA 052, a potential disease modifying anti-ILbeta antibody, shows sustained HbA1c reductions 3 months after a single injection with no increases in safety parameters in subjects with type 2 diabetes. Diabetes 58[Suppl. 1], A30. 2009. Ref Type: Abstract
- [Background] Rewers, A Klingensmith G Brown A Rewers M. Children presenting in DKA at diagnosis have higher HbA1cduring initial 8 years of type 1 diabetes independently of access to care and ethnicity. Pediatric Diabetes 8[Suppl. 7], 32. 2007. Ref Type: Abstract
- [Background] Glaser NS, Marcin JP, Wootton-Gorges SL, Buonocore MH, Rewers A, Strain J, DiCarlo J, Neely EK, Barnes P, Kuppermann N. Correlation of clinical and biochemical findings with diabetic ketoacidosis-related cerebral edema in children using magnetic resonance diffusion-weighted imaging. J Pediatr. 2008 Oct;153(4):541-6. doi: 10.1016/j.jpeds.2008.04.048. Epub 2008 Jun 27. PMID 18589447
- [Background] Quiros JA, Marcin JP, Kuppermann N, Nasrollahzadeh F, Rewers A, DiCarlo J, Neely EK, Glaser N. Elevated serum amylase and lipase in pediatric diabetic ketoacidosis. Pediatr Crit Care Med. 2008 Jul;9(4):418-22. doi: 10.1097/PCC.0b013e318172e99b. PMID 18496406
- [Background] Rewers A, McFann K, Chase HP. Bedside monitoring of blood beta-hydroxybutyrate levels in the management of diabetic ketoacidosis in children. Diabetes Technol Ther. 2006 Dec;8(6):671-6. doi: 10.1089/dia.2006.8.671. PMID 17109599
- [Background] Galea J, Ogungbenro K, Hulme S, Greenhalgh A, Aarons L, Scarth S, Hutchinson P, Grainger S, King A, Hopkins SJ, Rothwell N, Tyrrell P. Intravenous anakinra can achieve experimentally effective concentrations in the central nervous system within a therapeutic time window: results of a dose-ranging study. J Cereb Blood Flow Metab. 2011 Feb;31(2):439-47. doi: 10.1038/jcbfm.2010.103. Epub 2010 Jul 14. PMID 20628399
- [Background] Gueorguieva I, Clark SR, McMahon CJ, Scarth S, Rothwell NJ, Tyrrell PJ, Hopkins SJ, Rowland M. Pharmacokinetic modelling of interleukin-1 receptor antagonist in plasma and cerebrospinal fluid of patients following subarachnoid haemorrhage. Br J Clin Pharmacol. 2008 Mar;65(3):317-25. doi: 10.1111/j.1365-2125.2007.03026.x. Epub 2007 Sep 13. PMID 17875190
- [Background] DKA TREATMENT PROTOCOL Barbara Davis Center for Childhood Diabetes, University of Colorado & The Children's Hospital Denver. http://www.ucdenver.edu/academics/colleges/medicalschool/centers/BarbaraDavis/Pages/contact.aspx . 2010.
- [Background] Erlich H, Valdes AM, Noble J, Carlson JA, Varney M, Concannon P, Mychaleckyj JC, Todd JA, Bonella P, Fear AL, Lavant E, Louey A, Moonsamy P; Type 1 Diabetes Genetics Consortium. HLA DR-DQ haplotypes and genotypes and type 1 diabetes risk: analysis of the type 1 diabetes genetics consortium families. Diabetes. 2008 Apr;57(4):1084-92. doi: 10.2337/db07-1331. Epub 2008 Feb 5. PMID 18252895
- [Background] Soldatos T, Chatzimichail K, Papathanasiou M, Gouliamos A. Optic nerve sonography: a new window for the non-invasive evaluation of intracranial pressure in brain injury. Emerg Med J. 2009 Sep;26(9):630-4. doi: 10.1136/emj.2008.058453. PMID 19700575
- [Background] Karakitsos D, Soldatos T, Gouliamos A, Armaganidis A, Poularas J, Kalogeromitros A, Boletis J, Kostakis A, Karabinis A. Transorbital sonographic monitoring of optic nerve diameter in patients with severe brain injury. Transplant Proc. 2006 Dec;38(10):3700-6. doi: 10.1016/j.transproceed.2006.10.185. PMID 17175372
- [Background] Tayal VS, Neulander M, Norton HJ, Foster T, Saunders T, Blaivas M. Emergency department sonographic measurement of optic nerve sheath diameter to detect findings of increased intracranial pressure in adult head injury patients. Ann Emerg Med. 2007 Apr;49(4):508-14. doi: 10.1016/j.annemergmed.2006.06.040. Epub 2006 Sep 25. PMID 16997419
- [Background] Le A, Hoehn ME, Smith ME, Spentzas T, Schlappy D, Pershad J. Bedside sonographic measurement of optic nerve sheath diameter as a predictor of increased intracranial pressure in children. Ann Emerg Med. 2009 Jun;53(6):785-91. doi: 10.1016/j.annemergmed.2008.11.025. Epub 2009 Jan 23. PMID 19167786
- [Background] Auron PE, Webb AC, Rosenwasser LJ, Mucci SF, Rich A, Wolff SM, Dinarello CA. Nucleotide sequence of human monocyte interleukin 1 precursor cDNA. Proc Natl Acad Sci U S A. 1984 Dec;81(24):7907-11. doi: 10.1073/pnas.81.24.7907. PMID 6083565